CLINICAL TRIAL: NCT02776787
Title: DEBUT: Diverticulitis Evaluation of Patient Burden, Utilization, and Trajectory
Acronym: DEBUT
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Director, Surgical Outcomes Research Center, University of Washington
Other Study IDs: STUDY00003708; 1R01DK103915-01A1 (NIH)
Record Dates: First submitted 2016-05-05; First posted 2016-05-18 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with diverticulitis
- Surgeons: Surgeons who perform elective colon resections

SUMMARY:
Half of all Americans over 60 years of age have diverticulitis of the colon. Over the last decade, the use of elective colon resection has increased by more than 50%, and diverticulitis is now the leading reason for elective colectomy. Surgeons and patients alike have a difficult time deciding if surgery is the best choice to treat diverticulitis. The goal of the DEBUT study is to improve the understanding about how doctors and patients make decisions to have elective surgery for diverticulitis, and the global impact of diverticulitis on patients' lives.

DETAILED DESCRIPTION:
This study will examine both clinical and non-clinical reasons for pursuing surgery, taking into account previously unexplored areas in surgical decision-making including the comprehensive impact of this disease, as well as factors that impact a surgeon's willingness to recommend surgery. Ultimately, this patient-centered research approach will help us understand the impact of treatment decisions on a patient's quality of life, work, and clinical symptoms, and will ultimately help to inform our recommendations for the treatment of patients with diverticulitis.

The DEBUT study was developed from questions raised by our Washington State Surgical Collaborative, (SCOAP Colon and Rectal Surgery Work Group) and will be carried out in clinics and hospitals across Washington State, Oregon, and California. The investigators invite patients to participate in research activities designed to identify the impact of diverticulitis and treatment options, in order to better understand the outcomes that matter most to patients. Patients who are considering surgery or who have received treatment for their diverticulitis will be recruited for study participation. Participants will complete a baseline survey via a convenient electronic platform, and follow-up surveys will be sent quarterly for up to four years. These surveys will examine quality of life, overall health, and clinical symptoms to understand what drives patients and surgeons to an operation, as well as how that decision impacts quality of life and recurrent events in patients that choose to have surgery compared to those that do not have surgery. Participating surgeons will complete surveys that examine their indications for surgery and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of diverticulitis
* Patients 18 years of age or older
* Patients who are able to consent to participate in research

Exclusion Criteria:

* Patients that have had prior colon resection surgery
* Patients that do not make their own medical decisions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnoses of diverticulitis will be recruited from emergency rooms (first time episodes), GI clinics, and surgical clinics across the Pacific Northwest and California.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2016-03; Primary Completion 2021-01 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Patient-reported symptom burden and quality of life measured by the Diverticulitis Quality of Life scale (DV-QOL) | 3 months - 4 years
  Patient-reported burden of disease (diverticulitis symptoms and quality of life, as measured by the Diverticulitis Quality of Life scale (DV-QOL)) will be measured over time among patients that do and do not undergo elective colon resection.

SECONDARY OUTCOMES:
Number of patients who report non-clinical factors as reason for deciding to have surgery | 3 months - 4 years
  Patient-reported factors (clinical and non-clinical) for deciding to have elective colon surgery, or deciding to have medical management for diverticulitis will be analyzed across surgical and non-surgical patients.

CONTACTS AND LOCATIONS:
Overall Officials: Giana Davidson, MD, MPH, Study Director — University of Washington
Locations (9):
- United States (9):
  - UCLA Ronald Reagan, Los Angeles, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - NYU Langone Health, Brooklyn, New York
  - Legacy Health, Portland, Oregon
  - Skagit Regional Health, Mount Vernon, Washington
  - Valley Medical Center, Renton, Washington
  - Harborview Medical Center, Seattle, Washington
  - Northwest Hospital and Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No